CLINICAL TRIAL: NCT04883632
Title: A Prospective, Randomized, Multicenter Study Evaluating Saypha® VOLUME Lidocaine* for the Correction of Nasolabial Fold
Brief Title: Saypha® Volume LIdocaine in Nasolabial Folds
Acronym: SAVINO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Croma-Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPH-101-201477
Record Dates: First submitted 2021-05-11; First posted 2021-05-12 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-12

CONDITIONS: Moderate to Severe Nasolabial Folds

STUDY DESIGN:
Intervention Model Description: prospective, randomized, double-blind, parallel-group, multi-center study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomized to receive products from one of 2 productions sites. (C1 and HQ, respectively); as the products appear in an identical fashion only the batch numbers will allow identification of the production site; as the allocation of batch numbers to the respective site is not disclosed to the study site team, the entire team will be masked until break of blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volume Lidocaine HQ (Experimental): Subjects randomized to be treated with Saypha Volume Lidocaine manufactured in the Croma Pharma HQ Facility
  Interventions: Combination Product: Saypha Volume Lidocaine
- Volume Lidocaine C1 (Active Comparator): Subjects randomized to be treated with Saypha Volume Lidocaine manufactured in the Croma Pharma C1 Facility
  Interventions: Combination Product: Saypha Volume Lidocaine

INTERVENTIONS:
Combination Product: Saypha Volume Lidocaine — correction of Nasolabial Folds using injection of Saypha Volume Lidocaine manufactured in 2 different plants at Croma Pharma.
  The amount injected depended on the size of the area to be corrected and the desired level of soft tissue augmentation. It was estimated that a maximum volume of 4 mL per treatment was needed but should not have exceeded 10 mL in total per treatment or 20 mL per year. and use in respective indications. The investigational device was administered to eligible subjects on investigation Day 0. A touchup treatment at Week 2 was optional at the investigator's discretion if full correction was

SUMMARY:
Comparison of saypha Volume Lidocaine from 2 different manufacturing locations in correcting moderate to sever nasolabial folds

DETAILED DESCRIPTION:
Following informed consent and screening, eligible subjects with moderate to severe nasolabial folds will be randomized to receive saypha® VOLUME Lidocaine from 1 of 2 manufacturing sites. The device will be injected into the deep dermis or supraperiostal, and subjects will return for follow-up assessments at Week 2, 4, 24, 36, 52 and optional at Week 65, 78 and 104 after the treatment. A Touch-up treatment may be done at Week 2, if deemed appropriate by the investigator. The performance of the investigational device will be evaluated by the investigator by assessing severity of nasolabial folds using the Nasolabial Folds Severity Rating Scale (NLF-SRS) at Week 4, 24, 36, 52 after the treatment and optional at Week 65, 78 and 104 and in comparison to Day 0. Telephone visits will be performed approximately 24 hours post-administration to monitor possible adverse events. In case any adverse events are reported during the telephone visits an unscheduled visit should be performed.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet ALL of the following criteria to be eligible for the study:

1. Male or female 18 years of age or older
2. Presence of two fully visible, approximately symmetrical nasolabial folds, with each of the folds scored with 2 or 3 according to the 5-grade Nasolabial Folds Severity Rating Scale (NLF-SRS) as assessed by the investigator
3. Healthy skin in the facial area and free of diseases that could interfere in cutaneous aging evaluation
4. Willingness to abstain from any aesthetic or surgical procedures in the treatment area for the duration of the clinical investigation
5. Written signed and dated informed consent

Exclusion Criteria:

subject who meets ANY of the following criteria is NOT eligible for the study:

1. Pregnancy, lactation, planned pregnancy or unwillingness to use contraception at any time during the study (for women of child-bearing potential only)
2. History of mental disorders or emotional instability
3. History of allergic reaction or hypersensitivity to hyaluronic acid, lidocaine, or any amide-based anaesthetic
4. Presence of silicone implant or another non-absorbable substance (permanent fillers) in the nasolabial region
5. Any superficial or deep facial surgery or injection or implantation of any dermal fillers (including but not limited to hyaluronic acid, collagen, calcium hydroxylapatite, poly-l-lactic acid, polymethylmethacrylate, autologous fat injections), application of any absorbable and non-absorbable sutures (thread) for any purpose including wound care and facial lifting, any laser therapy (including but not limited to Neodym-YAG, KTP, IPL, Diode lasers as well as Erbium-YAG, CO2 or other ablative lasers), dermoabrasion, or botulinum toxin application in the nasolabial region within previous 12 months prior to enrolment, or any chemical peeling procedures (including but not limited to glycolic acid, trichloroacetic acid or phenolic peels) within previous 3 months prior to enrolment, or planning to undergo such procedures in the treatment area during the study
6. Presence of infectious, inflammatory, or proliferative lesions in the nasolabial region
7. Cutaneous lesions in the treatment area
8. Known human immune deficiency virus-positive individuals
9. History of allergies against aesthetic filling products and recurrent (3 times a year) herpes simplex in the treated area
10. Tendency to hypertrophic scars and/or keloid formation
11. History or presence of any autoimmune or connective tissue disease, or current treatment with immune therapy
12. Uncontrolled systemic diseases (such as diabetes mellitus)
13. Bariatric surgery within 12 months prior to enrollment or planned during the clinical investigation
14. Use of anticoagulant or thrombolytic medication from 10 days pre- to 3 days post injection
15. Any medical condition which, in the investigator's opinion, prohibits the inclusion in the study
16. Current or previous (within 30 days of enrolment) treatment with another investigational drug and/or medical device or participation in another clinical study
17. Previous enrolment in this clinical investigation
18. Subjects whose participation in clinical trials is prohibited by the Austrian Medical Devices Act (e.g., persons with a legal custodian appointed due to mental disability, prisoners, soldiers and other members of the armed forces, civil servants)
19. Any dental procedures one month before until one month after treatment with the investigational device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Austria (3):
  - Yuvell, Vienna
  - Ordination Dr. Gaerner, Vienna
  - Privatklinik Waehring GmbH, Vienna

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment:110 (Subjects enrolled include subjects screened and randomized))
Groups:
- Saypha® VOLUME Lidocaine HQ: Subjects who had administration of saypha® VOLUME Lidocaine manufactured in HQ
- Saypha® VOLUME Lidocaine C1: Subjects who had administation of Sapha® VOLUME manufactured in C1
Period: Overall Study
Arm/Group | Saypha® VOLUME Lidocaine HQ | Saypha® VOLUME Lidocaine C1
Started | 55 | 55
Completed | 53 | 52
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Population: The data sets contain all data collected in the Intent-to-treat population (ITT), which is defined as all subjects who received the investigational device and have at least one post-treatment assessment N =109 The SAF (Safety analysis Set) also has N = 109 Number of subjects with trial completion at week 24: N =106
Groups:
- Volume Lidocaine HQ: Subjects randomized to be treated with Saypha Volume Lidocaine manufactured in the Croma Pharma HQ Facility
  Saypha Volume Lidocaine: correction of Nasolabial Folds using injection of Saypha Volume Lidocaine manufactured in 2 different plants at Croma Pharma
- Volume Lidocaine C1: Subjects randomized to be treated with Saypha Volume Lidocaine manufactured in the Croma Pharma C1 Facility
  Saypha Volume Lidocaine: correction of Nasolabial Folds using injection of Saypha Volume Lidocaine manufactured in 2 different plants at Croma Pharma
- Total: Total of all reporting groups
Arm/Group | Volume Lidocaine HQ | Volume Lidocaine C1 | Total
Number analyzed (Participants) | 54 | 55 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (10.1) | 48.8 (7.9) | 49.2 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 50 | 102
  Male | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 52 | 53 | 105
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Nasolabial fold severity scale - Grading by investigator [Count of Participants; unit: Participants]
  left side: 0 = None/minimal | 0 | 0 | 0
  left side: 1 = Mild | 0 | 0 | 0
  left side: 2 = Moderate | 27 | 30 | 57
  left side: 3 = Severe | 27 | 25 | 52
  left side: 4 = Extreme | 0 | 0 | 0
  right side: 0 = None/minimal | 0 | 0 | 0
  right side: 1 = Mild | 0 | 0 | 0
  right side: 2 = Moderate | 33 | 32 | 65
  right side: 3 = Severe | 21 | 23 | 44
  right side: 4 = Extreme | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate in Reduction of Nasolabial Folds
Description: The proportion of subjects with the NLF-SRS grade reduced by ≥1 point versus baseline at Week 24. This anaylsis is done per manufacturing site: C1 and HQ separately and for the overall population. A 'responder' is defined having at least ≥ 1 grade improvement as evaluated with the 5 point-validated NLF-SRS score on both sides of the face.
  Nasolabial Folds Severity Rating Scale (NLF-SRS) is a validated 5 grade scale where the lower number corresponds to:
  0 = None/minimal: No visible/minimal nasolabial folds;
  1. = Mild: Shallow but visible nasolabial fold with a slight indentation;
  2. = Moderate: Moderately deep nasolabial fold;
  3. = Severe: Very deep nasolabial fold with prominent facial feature;
  4. = Extreme: Extremely deep and long nasolabial fold with skin redundancy
  Therefore, the lower the number, the better.
Time Frame: 24 Weeks
Population: The primary data set for analyses of performance of the investigational device and of aesthetic effects will contain all data collected in the Intent-to-treat population, which is defined as all subjects who received the investigational device and have at least one post-treatment assessment, but for this analysis we have to consider the number of subjects with trial completion at Week 24, threfore an overal population of 106.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Population (Saypha Volume Lidocaine HQ + C1): Subjects randomized to be treated with Saypha Volume Lidocaine manufactured in both facilities
Arm/Group | Volume Lidocaine HQ | Volume Lidocaine C1 | Overall Population (Saypha Volume Lidocaine HQ + C1)
Number analyzed (Participants) | 53 | 53 | 106
Participants | 34 | 39 | 73

2. Secondary Outcome: Proportion of Responders at Other Time Points
Description: The proportion of subjects with the NLF-SRS grade reduced by ≥1 point versus baseline at Week 4, Week 36, Week 52 and optional at Week 65, Week 78 and Week 104.
  A reduction in the score of the Nasolabial Folds Severity Rating Scale is considered an improvement as this reflects a decrease of the folds severity which is rated from 0 (none/minimal) to 4 (extreme).
  Individual NLF-SRS grades per visit calculated as the mean of grades assigned to the left and the right NLF, respectively
  On the Nasolabial Fold-Severity Rating Scale (NLF-SRS) higher scores indicate a greater severity of the folds: 0 = None/minimal: No visible/minimal nasolabial folds, 1 = Mild: Shallow but visible nasolabial fold with a slight indentation, 2 = Moderate: Moderately deep nasolabial fold, 3 = Severe: Very deep nasolabial fold with prominent facial feature, 4 = Extreme: Extremely deep and long nasolabial fold with skin redundancy
Time Frame: Week 4, week 36, week 52, week 65, week 78, week 104
Population: The primary data set for analyses of performance of the investigational device and of aesthetic effects will contain all data collected in the Intent-to-treat population, which is defined as all subjects who received the investigational device and have at least one post-treatment assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Volume Lidocaine HQ | Volume Lidocaine C1 | Overall Population (Saypha Volume Lidocaine HQ + C1)
Number analyzed (Participants) | 54 | 55 | 109
Participants
  Week 4: number analyzed (Participants) | 50 | 50 | 100
  Week 4 | 46 | 46 | 92
  Week 36: number analyzed (Participants) | 53 | 53 | 106
  Week 36 | 27 | 32 | 59
  Week 52: number analyzed (Participants) | 53 | 52 | 105
  Week 52 | 10 | 13 | 23
  Week 65: number analyzed (Participants) | 13 | 16 | 29
  Week 65 | 3 | 3 | 6
  Week 78: number analyzed (Participants) | 6 | 5 | 11
  Week 78 | 1 | 0 | 1
  Week 104: number analyzed (Participants) | 1 | 0 | 1
  Week 104 | 0 | 0 | 0

3. Secondary Outcome: Change Versus Baseline in Nasolabial Fold Severitry
Description: The average change versus baseline in the NLF-SRS (Nasolabial Folds Severity Rating Scale) grade at Week 4, Week 24, Week 36, Week 52 and, optional at Week 65, Week 78 and Week 104 as evaluated by the investigator.
  A reduction in the score of the Nasolabial Folds Severity Rating Scale is considered an improvement as this reflects a decrease of the folds severity which is rated from 0 (none/minimal) to 4 (extreme).
  Nasolabial Folds Severity Rating Scale (NLF-SRS) is a validated 5 grade scale where the lower number corresponds to:
  0 = None/minimal: No visible/minimal nasolabial folds;
  1. = Mild: Shallow but visible nasolabial fold with a slight indentation;
  2. = Moderate: Moderately deep nasolabial fold;
  3. = Severe: Very deep nasolabial fold with prominent facial feature;
  4. = Extreme: Extremely deep and long nasolabial fold with skin redundancy
  Therefore, the lower the number, the better.
Time Frame: Week 4, Week 24, Week 36, Week 52 and, optional at Week 65, Week 78 and Week 104
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Volume Lidocaine HQ | Volume Lidocaine C1 | Overall Population (Saypha Volume Lidocaine HQ + C1)
Number analyzed (Participants) | 54 | 55 | 109
score on a scale
  Week 4: number analyzed (Participants) | 50 | 50 | 100
  Week 4 | 1.4 (0.6) | 1.4 (0.6) | 1.4 (0.6)
  Week 24: number analyzed (Participants) | 53 | 53 | 106
  Week 24 | 1.0 (0.90) | 1.2 (0.80) | 1.1 (0.90)
  Week 36: number analyzed (Participants) | 53 | 53 | 106
  Week 36 | 0.7 (0.8) | 0.7 (0.7) | 0.7 (0.8)
  Week 52: number analyzed (Participants) | 53 | 52 | 105
  Week 52 | 0.2 (0.5) | 0.3 (0.5) | 0.2 (0.5)
  Week 65: number analyzed (Participants) | 13 | 16 | 29
  Week 65 | 0.2 (0.7) | 0.1 (0.6) | 0.1 (0.6)
  Week 78: number analyzed (Participants) | 6 | 5 | 11
  Week 78 | 0.3 (0.5) | 0.0 (0.7) | 0.2 (0.6)
  Week 104: number analyzed (Participants) | 1 | 0 | 1
  Week 104 | 0.0 |  | 0.0

4. Other Pre Specified Outcome: Percentage of Responders With a ≥2-point Improvement
Description: Percentage of responders with a ≥2-point improvement over Baseline on the 5-point NLF-SRS, based on investigator's live assessment at Weeks 4, 24, 36, 52, 65, 78, and 104 after initial treatment.
  On the Nasolabial Fold-Severity Rating Scale (NLF-SRS) higher scores indicate a greater severity of the folds: 0 = None/minimal: No visible/minimal nasolabial folds, 1 = Mild: Shallow but visible nasolabial fold with a slight indentation, 2 = Moderate: Moderately deep nasolabial fold, 3 = Severe: Very deep nasolabial fold with prominent facial feature, 4 = Extreme: Extremely deep and long nasolabial fold with skin redundancy
Time Frame: Weeks 4, 24, 36, 52, 65, 78, and 104
Population: The primary data set for analyses of performance of the investigational device and of aesthetic effects will contain all data collected in the Intent-to-treat population, which is defined as all subjects who received the investigational device and have at least one post-treatment assessment. In the protocol and statistical analysis plan, the analysis for this outcome measure was planned only for the overall population and not for the randomized subgroups.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Population (Saypha Volume Lidocaine HQ + C1): Subjects randomized to be treated with Saypha Volume Lidocaine in total
  Saypha Volume Lidocaine: correction of Nasolabial Folds using injection of Saypha Volume Lidocaine manufactured in 2 different plants at Croma Pharma
Arm/Group | Overall Population (Saypha Volume Lidocaine HQ + C1)
Number analyzed (Participants) | 109
Participants
  Week 4: number analyzed (Participants) | 100
  Week 4 | 43
  Week 24: number analyzed (Participants) | 106
  Week 24 | 32
  Week 36: number analyzed (Participants) | 106
  Week 36 | 12
  Week 52: number analyzed (Participants) | 105
  Week 52 | 0
  Week 65: number analyzed (Participants) | 29
  Week 65 | 0
  Week 78: number analyzed (Participants) | 11
  Week 78 | 0
  Week 104: number analyzed (Participants) | 1
  Week 104 | 0

5. Other Pre Specified Outcome: Percentage of Subjects With Aesthetic Improvement Using the 5-point GAIS Based on Investigator's Assessment
Description: Percentage of subjects with aesthetic improvement using the 5-point Global Aesthetzic Improvement Scavel (GAIS) (subjects who have been rated as "very much improved" or "much improved" or "improved"), based on investigator's assessment at Weeks 4, 24, 36, 52, 65, 78, and 104 after initial treatment, for each treatment location (right NLF, left NLF) separately and overall.
Time Frame: Weeks 4, 24, 36, 52, 65, 78, and 104
Population: The primary data set for analyses of performance of the investigational device and of aesthetic effects will contain all data collected in the Intent-to-treat population, which is defined as all subjects who received the investigational device and have at least one post-treatment assessment. In the protocol and statistical analysis plan, the analysis for this outcome measure was planned only for the overall population and not for the randomized subgroups Saypha® FILLER HQ and Saypha® FILLER C1
Measure: Count of Participants; unit: Participants
Groups:
- Overall Population (Saypha Volume Lidocaine HQ + C1) - Left Nasolabial Fold: Subjects randomized to be treated with Saypha Volume Lidocaine in total
  Saypha Volume Lidocaine: correction of Nasolabial Folds using injection of Saypha Volume Lidocaine manufactured in 2 different plants at Croma Pharma
  GAIS Improvement rates by Investigator for left Nasolabial Fold
- Overall Population (Saypha Volume Lidocaine HQ + C1) - Right Nasolabial Fold: Subjects randomized to be treated with Saypha Volume Lidocaine in total
  Saypha Volume Lidocaine: correction of Nasolabial Folds using injection of Saypha Volume Lidocaine manufactured in 2 different plants at Croma Pharma
  GAIS Improvement rates by Investigator for right Nasolabial Fold
- Overall Population (Saypha Volume Lidocaine HQ + C1) - Volume Lidocaine: Subjects randomized to be treated with Saypha Volume Lidocaine in total
  Saypha Volume Lidocaine: correction of Nasolabial Folds using injection of Saypha Volume Lidocaine manufactured in 2 different plants at Croma Pharma
  Improvement Rates by Investigator in both treatment locations (left and right Nasolabialfold)
Arm/Group | Overall Population (Saypha Volume Lidocaine HQ + C1) - Left Nasolabial Fold | Overall Population (Saypha Volume Lidocaine HQ + C1) - Right Nasolabial Fold | Overall Population (Saypha Volume Lidocaine HQ + C1) - Volume Lidocaine
Number analyzed (Participants) | 109 | 109 | 109
Participants
  Week 4: number analyzed (Participants) | 100 | 100 | 100
  Week 4: No Improvement | 0 | 2 | 2
  Week 4: Improvement | 100 | 98 | 98
  Week 24: number analyzed (Participants) | 106 | 106 | 106
  Week 24: No Improvement | 17 | 16 | 18
  Week 24: Improvement | 89 | 90 | 88
  Week 36: number analyzed (Participants) | 106 | 106 | 106
  Week 36: No Improvement | 44 | 43 | 45
  Week 36: Improvement | 62 | 63 | 61
  Week 52: number analyzed (Participants) | 105 | 105 | 105
  Week 52: No Improvement | 76 | 73 | 76
  Week 52: Improvement | 29 | 32 | 29
  Week 65: number analyzed (Participants) | 29 | 29 | 29
  Week 65: No Improvement | 19 | 20 | 20
  Week 65: Improvement | 10 | 9 | 9
  Week 78: number analyzed (Participants) | 11 | 11 | 11
  Week 78: No Improvement | 10 | 10 | 10
  Week 78: Improvement | 1 | 1 | 1
  Week 104: number analyzed (Participants) | 1 | 1 | 1
  Week 104: No Improvement | 1 | 1 | 1
  Week 104: Improvement | 0 | 0 | 0

6. Other Pre Specified Outcome: Percentage of Subjects With Aesthetic Improvement Using the 5-point GAIS Based on Subjects Assessment
Description: Percentage of subjects with aesthetic improvement using the 5-point Global Aesthetzic Improvement Scavel (GAIS) (subjects who have been rated as "very much improved" or "much improved" or "improved"), based on subject's assessment at Weeks 4, 24, 36, 52, 65, 78, and 104 after initial treatment, for each treatment location (right NLF, left NLF) separately and overall.
Time Frame: Weeks 4, 24, 36, 52, 65, 78, and 104
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Groups:
- Overall Population (Saypha Volume Lidocaine HQ + C1) - Left Nasolabial Fold: Subjects randomized to be treated with Saypha Volume Lidocaine in total
  Saypha Volume Lidocaine: correction of Nasolabial Folds using injection of Saypha Volume Lidocaine manufactured in 2 different plants at Croma Pharma
  GAIS Improvement rates by subject for left Nasolabial Fold
- Overall Population (Saypha Volume Lidocaine HQ + C1) - Right Nasolabial Fold: Subjects randomized to be treated with Saypha Volume Lidocaine in total
  Saypha Volume Lidocaine: correction of Nasolabial Folds using injection of Saypha Volume Lidocaine manufactured in 2 different plants at Croma Pharma
  GAIS Improvement rates by subject for right Nasolabial Fold
- Overall Population (Saypha Volume Lidocaine HQ + C1) - Volume Lidocaine: Subjects randomized to be treated with Saypha Volume Lidocaine in total
  Saypha Volume Lidocaine: correction of Nasolabial Folds using injection of Saypha Volume Lidocaine manufactured in 2 different plants at Croma Pharma
  Improvement Rates by subject in both treatment locations (left and right Nasolabialfold)
Arm/Group | Overall Population (Saypha Volume Lidocaine HQ + C1) - Left Nasolabial Fold | Overall Population (Saypha Volume Lidocaine HQ + C1) - Right Nasolabial Fold | Overall Population (Saypha Volume Lidocaine HQ + C1) - Volume Lidocaine
Number analyzed (Participants) | 109 | 109 | 109
Participants
  Week 4: number analyzed (Participants) | 106 | 106 | 106
  Week 4: No improvement | 3 | 2 | 3
  Week 4: Improvement | 103 | 104 | 103
  Week 24: number analyzed (Participants) | 107 | 107 | 107
  Week 24: No improvement | 12 | 13 | 13
  Week 24: Improvement | 95 | 94 | 94
  Week 36: number analyzed (Participants) | 106 | 106 | 106
  Week 36: No improvement | 26 | 22 | 26
  Week 36: Improvement | 80 | 84 | 80
  Week 52: number analyzed (Participants) | 105 | 105 | 105
  Week 52: No improvement | 51 | 49 | 51
  Week 52: Improvement | 54 | 56 | 54
  Week 65: number analyzed (Participants) | 29 | 29 | 29
  Week 65: No improvement | 17 | 17 | 17
  Week 65: Improvement | 12 | 12 | 12
  Week 78: number analyzed (Participants) | 11 | 11 | 11
  Week 78: No improvement | 6 | 6 | 6
  Week 78: Improvement | 5 | 5 | 5
  Week 104: number analyzed (Participants) | 1 | 1 | 1
  Week 104: No improvement | 1 | 1 | 1
  Week 104: Improvement | 0 | 0 | 0

7. Other Pre Specified Outcome: Percentage of Responders With a ≥1-point Improvement Over Baseline on the 5-point NLF-SRS, Based on Evaluation by an Independent Reviewer of Photographs
Description: Percentage of responders with a ≥1-point improvement over Baseline on the 5-point NLF-SRS, based on evaluation by an independent reviewer of photographs for Weeks 4, 36, 52, 65, 78, and 104 after initial treatment.
  On the Nasolabial Fold-Severity Rating Scale (NLF-SRS) higher scores indicate a greater severity of the folds: 0 = None/minimal: No visible/minimal nasolabial folds, 1 = Mild: Shallow but visible nasolabial fold with a slight indentation, 2 = Moderate: Moderately deep nasolabial fold, 3 = Severe: Very deep nasolabial fold with prominent facial feature, 4 = Extreme: Extremely deep and long nasolabial fold with skin redundancy
Time Frame: Weeks 4, 36, 52, 65, 78, and 104
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Population (Saypha Volume Lidocaine HQ + C1)
Number analyzed (Participants) | 109
Participants
  Week 4 : Response Rate with improvement 1 grade: number analyzed (Participants) | 100
  Week 4 : Response Rate with improvement 1 grade | 24
  Week 4 : Response Rate with improvement 2 grades: number analyzed (Participants) | 100
  Week 4 : Response Rate with improvement 2 grades | 3
  Week 24 : Response Rate with improvement 1 grade: number analyzed (Participants) | 106
  Week 24 : Response Rate with improvement 1 grade | 24
  Week 24 : Response Rate with improvement 2 grades: number analyzed (Participants) | 106
  Week 24 : Response Rate with improvement 2 grades | 0
  Week 36 : Response Rate with improvement 1 grade: number analyzed (Participants) | 106
  Week 36 : Response Rate with improvement 1 grade | 21
  Week 36 : Response Rate with improvement 2 grades: number analyzed (Participants) | 106
  Week 36 : Response Rate with improvement 2 grades | 0
  Week 52 : Response Rate with improvement 1 grade: number analyzed (Participants) | 104
  Week 52 : Response Rate with improvement 1 grade | 19
  Week 52 : Response Rate with improvement 2 grades: number analyzed (Participants) | 104
  Week 52 : Response Rate with improvement 2 grades | 1
  Week 65 : Response Rate with improvement 1 grade: number analyzed (Participants) | 29
  Week 65 : Response Rate with improvement 1 grade | 8
  Week 65 : Response Rate with improvement 2 grades: number analyzed (Participants) | 29
  Week 65 : Response Rate with improvement 2 grades | 1
  Week 78 : Response Rate with improvement 1 grade: number analyzed (Participants) | 11
  Week 78 : Response Rate with improvement 1 grade | 4
  Week 78 : Response Rate with improvement 2 grades: number analyzed (Participants) | 11
  Week 78 : Response Rate with improvement 2 grades | 0
  Week 104 : Response Rate with improvement 1 grade: number analyzed (Participants) | 1
  Week 104 : Response Rate with improvement 1 grade | 1
  Week 104 : Response Rate with improvement 2 grades: number analyzed (Participants) | 1
  Week 104 : Response Rate with improvement 2 grades | 0

8. Other Pre Specified Outcome: Subject Satisfaction With Outcome of the Treatment, Assessed by the Face-Q Questionnaire "Satisfaction With Outcome"
Description: Descriptive summary statistics for extent of subject satisfaction with outcome of the treatment, as assessed by the Face-Q questionnaire "Satisfaction with Outcome" at Weeks 4, 24, 36, 52, 65, 78, and 104 after initial treatment.
  Face-Q TM Questionnaire "Satisfaction with Outcome", a 6- tem, Health-related Quality of Life Questionnaire: The raw summed scale score is converted to a score from 0 to 100 by using the transformed sum score (Rasch model): Modified sum score ranges from 0 to 100 (low numbers correspond to low satisfaction).
Time Frame: Weeks 4, 24, 36, 52, 65, 78, and 104
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Overall Population (Saypha Volume Lidocaine HQ + C1)
Number analyzed (Participants) | 109
score on a scale
  Week 4: number analyzed (Participants) | 106
  Week 4 | 76.8 (18.9)
  Week 24: number analyzed (Participants) | 107
  Week 24 | 71.1 (23.7)
  Week 36: number analyzed (Participants) | 106
  Week 36 | 62.2 (25.3)
  Week 52: number analyzed (Participants) | 105
  Week 52 | 60.1 (27.9)
  Week 65: number analyzed (Participants) | 29
  Week 65 | 83.9 (18.0)
  Week 78: number analyzed (Participants) | 11
  Week 78 | 77.4 (23.1)
  Week 104: number analyzed (Participants) | 1
  Week 104 | 59.0

9. Other Pre Specified Outcome: Pain Intensity, as Evaluated by the Subject Using an 11-point NPRS
Description: Descriptive summary statistics for pain intensity, as evaluated by the subject using an 11-point NPRS (where 0 is no pain and 10 is the worst pain imaginable) immediately after the last injection and 15 minutes thereafter, at Day 0 and optional at Week 2.
Time Frame: Day 0 and Week 2.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Population (Saypha Volume Lidocaine HQ + C1)
Number analyzed (Participants) | 109
units on a scale
  Injection at Day 0 - immediately after injection | 1.4 (1.4)
  Injection at Day 0 - 15 minutes after injection | 0.0 (0.2)
  Injection at Week 2 - immediately after injection: number analyzed (Participants) | 26
  Injection at Week 2 - immediately after injection | 0.8 (1.1)
  Injection at Week 2 - 15 minutes after injection: number analyzed (Participants) | 25
  Injection at Week 2 - 15 minutes after injection | 0.0 (0.0)

10. Other Pre Specified Outcome: Percentage of Subjects Having an Aesthetic Effect
Description: Percentage of subjects having an aesthetic effect, based on the investigator's life assessment at Weeks 24, 36, 52, 65, 78, and 104.
Time Frame: Weeks 24, 36, 52, 65, 78, and 104
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Volume Lidocaine HQ | Volume Lidocaine C1 | Overall Population (Saypha Volume Lidocaine HQ + C1)
Number analyzed (Participants) | 53 | 54 | 107
Participants
  Week 24: number analyzed (Participants) | 53 | 53 | 106
  Week 24: Aesthetic effect still present - yes | 43 | 47 | 90
  Week 24: Aesthetic effect still present - no | 10 | 6 | 16
  Week 36: number analyzed (Participants) | 53 | 53 | 106
  Week 36: Aesthetic effect still present - yes | 30 | 35 | 65
  Week 36: Aesthetic effect still present - no | 23 | 18 | 41
  Week 52: number analyzed (Participants) | 53 | 52 | 105
  Week 52: Aesthetic effect still present - yes | 14 | 17 | 31
  Week 52: Aesthetic effect still present - no | 39 | 35 | 74
  Week 65: number analyzed (Participants) | 13 | 16 | 29
  Week 65: Aesthetic effect still present - yes | 5 | 5 | 10
  Week 65: Aesthetic effect still present - no | 8 | 11 | 19
  Week 78: number analyzed (Participants) | 6 | 5 | 11
  Week 78: Aesthetic effect still present - yes | 1 | 0 | 1
  Week 78: Aesthetic effect still present - no | 5 | 5 | 10
  Week 104: number analyzed (Participants) | 1 | 0 | 1
  Week 104: Aesthetic effect still present - yes | 0 | 0 | 0
  Week 104: Aesthetic effect still present - no | 1 | 0 | 1

11. Other Pre Specified Outcome: The Proportion of Subjects With the NLF-SRS Grade Reduced by ≥1 Point Versus Baseline by Injection Technique and Device
Description: The proportion of subjects with the NLF-SRS grade reduced by ≥1 point versus Baseline at Weeks 4, 24, 36, 52, 65, 78, and 104 by injection technique (retrograde, bolus) and device (needle, cannula).
  A reduction in the score of the Nasolabial Folds Severity Rating Scale is considered an improvement as this reflects a decrease of the folds severity which is rated from 0 (none/minimal) to 4 (extreme).
  Nasolabial Folds Severity Rating Scale (NLF-SRS) is a validated 5 grade scale where the lower number corresponds to:
  0 = None/minimal: No visible/minimal nasolabial folds;
  1. = Mild: Shallow but visible nasolabial fold with a slight indentation;
  2. = Moderate: Moderately deep nasolabial fold;
  3. = Severe: Very deep nasolabial fold with prominent facial feature;
  4. = Extreme: Extremely deep and long nasolabial fold with skin redundancy
  Therefore, the lower the number, the better.
Time Frame: Week 4, Week 24, Week 36, Week 52 and, optional at Week 65, Week 78 and Week 104
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Subgroup 'Retrograde Technique': Subjects randomized to be treated with Saypha Volume Lidocaine The investigational device was administered with retrograde technique
- Subgroup "Bolus Technique": Subjects randomized to be treated with Saypha Volume Lidocaine The investigational device was administered with bolus technique
- Subgroup "Needle": Subjects randomized to be treated with Saypha Volume Lidocaine The investigational device was administered with a needle
- Subgroup "Cannula": Subjects randomized to be treated with Saypha Volume Lidocaine The investigational device was administered with a cannula
Arm/Group | Subgroup 'Retrograde Technique' | Subgroup "Bolus Technique" | Subgroup "Needle" | Subgroup "Cannula"
Number analyzed (Participants) | 58 | 51 | 63 | 46
Participants
  Week 4 after initial treatment: number analyzed (Participants) | 53 | 47 | 56 | 44
  Week 4 after initial treatment | 50 | 42 | 50 | 42
  Week 24 after initial treatment: number analyzed (Participants) | 57 | 49 | 61 | 45
  Week 24 after initial treatment | 40 | 33 | 40 | 33
  Week 36 after initial treatment: number analyzed (Participants) | 56 | 50 | 61 | 45
  Week 36 after initial treatment | 36 | 23 | 29 | 30
  Week 52 after initial treatment: number analyzed (Participants) | 55 | 50 | 61 | 44
  Week 52 after initial treatment | 13 | 10 | 15 | 8
  Week 65 after initial treatment: number analyzed (Participants) | 17 | 12 | 17 | 12
  Week 65 after initial treatment | 2 | 4 | 5 | 1
  Week 78 after initial treatment: number analyzed (Participants) | 5 | 6 | 8 | 3
  Week 78 after initial treatment | 1 | 0 | 1 | 0
  Week 104 after initial treatment: number analyzed (Participants) | 1 | 0 | 1 | 0
  Week 104 after initial treatment | 0 | 0 | 0 | 0

12. Other Pre Specified Outcome: Average Change Versus Baseline in the NLF-SRS Grade at Week 4, 24, 36, 52, 65, 78, and 104 as Evaluated by the Investigator by Injection Technique ('Retrograde', 'Bolus') and Device ('Needle', 'Cannula')
Description: The average change versus Baseline in the NLF-SRS grade at Weeks 4, 24, 36, 52, 65, 78, and 104 as evaluated by the investigator by injection technique ('retrograde', 'bolus') and device ('needle', 'cannula')
  On the Nasolabial Fold-Severity Rating Scale (NLF-SRS) higher scores indicate a greater severity of the folds: 0 = None/minimal: No visible/minimal nasolabial folds, 1 = Mild: Shallow but visible nasolabial fold with a slight indentation, 2 = Moderate: Moderately deep nasolabial fold, 3 = Severe: Very deep nasolabial fold with prominent facial feature, 4 = Extreme: Extremely deep and long nasolabial fold with skin redundancy
Time Frame: Week 4, 24, 36, 52, 65, 78, and 104
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subgroup 'Retrograde Technique' | Subgroup "Bolus Technique" | Subgroup "Needle" | Subgroup "Cannula"
Number analyzed (Participants) | 58 | 51 | 63 | 46
score on a scale
  Week 4: number analyzed (Participants) | 53 | 47 | 56 | 44
  Week 4 | 1.5 (0.5) | 1.3 (0.7) | 1.4 (0.6) | 1.5 (0.5)
  Week 24: number analyzed (Participants) | 57 | 49 | 61 | 45
  Week 24 | 1.1 (0.9) | 1.0 (0.9) | 1.0 (0.8) | 1.2 (0.9)
  Week 36: number analyzed (Participants) | 56 | 50 | 61 | 45
  Week 36 | 0.8 (0.7) | 0.6 (0.8) | 0.6 (0.8) | 0.9 (0.7)
  Week 52: number analyzed (Participants) | 55 | 50 | 61 | 44
  Week 52 | 0.3 (0.5) | 0.2 (0.5) | 0.2 (0.5) | 0.3 (0.4)
  Week 65: number analyzed (Participants) | 17 | 12 | 17 | 12
  Week 65 | 0.1 (0.6) | 0.3 (0.8) | 0.2 (0.7) | 0.0 (0.6)
  Week 78: number analyzed (Participants) | 5 | 6 | 8 | 3
  Week 78 | 0.2 (0.8) | 0.2 (0.4) | 0.3 (0.7) | 0.0 (0.0)
  Week 104: number analyzed (Participants) | 1 | 0 | 1 | 0
  Week 104 | 0.0 |  | 0.0 |

13. Other Pre Specified Outcome: Safety Outcome
Description: Occurrence and frequency of adverse events within each manufacturing site - HQ and C1 separately and for the overall population (HQ +C1). The safety of the investigational device will be monitored throughout the investigation, from visit 1 (Day 0 - baseline / treatment) until the final visit ( week 65 / visit 9). AEs were collected at each visit. In addition, the subjects were instructed to immediately contact the investigator by phone in case of occurrence of any untoward event between the visits.-
Time Frame: Day 0 until week 65
Population: All safety analyses will be based on the safety analysis set, defined as all subjects who received the investigational device (109 subjects). TEAEs is defined as treatment-emergent adverse event, that can be local and non local. Local TEAEs are the AEs in treatment area or just around treatment area; Non-Local: are AEs accredited to an IMD dose, if the start of AE is at the time point of application or later. In the below data local and non-local are reported together under TEAEs.
Measure: Count of Participants; unit: Participants
Arm/Group | Volume Lidocaine HQ | Volume Lidocaine C1 | Overall Population (Saypha Volume Lidocaine HQ + C1)
Number analyzed (Participants) | 54 | 55 | 109
Participants
  TEAES (local) - number of AEs reported | 11 | 4 | 15
  TEAES ( non-local) - number of AEs reported | 10 | 14 | 24
  TEAES (local)- Causal Relationship with IMP (probable + definite) | 6 | 4 | 10
  TEAES (non-local)- Causal Relationship with IMP (probable + definite) | 0 | 0 | 0
  TEAES (local) - Causal Relationship with Procedure (probable + definite) | 8 | 4 | 12
  TEAES (non-local) - Causal Relationship with Procedure (probable + definite) | 0 | 0 | 0
  TEAES (local) - SAEs | 0 | 0 | 0
  TEAES (non -local) - SAEs | 1 | 2 | 3

ADVERSE EVENTS:
Time Frame: 65 weeks. From day 0 ( IMP administration) until visit 9 ( week 65).
Description: AEs will be detected at each visit by clinical examination and by asking the subject about the occurrence of AEs. Care should be taken not to introduce bias when eliciting AE information from the subject.In addition, the subjects will be instructed to immediately contact the investigator/study site in case of occurrence of any untoward event between visits.
Arm/Group | Volume Lidocaine HQ | Volume Lidocaine C1 | Overall Population (Saypha Volume Lidocaine HQ + C1)
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/55 | 0/109
Serious Adverse Events (participants affected / at risk) | 1/54 | 2/55 | 3/109
Other Adverse Events (participants affected / at risk) | 16/54 | 14/55 | 30/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Volume Lidocaine HQ (N=54) | Volume Lidocaine C1 (N=55) | Overall Population (Saypha Volume Lidocaine HQ + C1) (N=109)
intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
vertebral foraminal stenosis, (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Volume Lidocaine HQ (N=54) | Volume Lidocaine C1 (N=55) | Overall Population (Saypha Volume Lidocaine HQ + C1) (N=109)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Administration site haematoma (General disorders) | 0 (0) | 1 (1) | 1 (1)
Administration site pain (General disorders) | 4 (4) | 0 (0) | 4 (4)
Administration Site swelling (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection Site Pain (General disorders) | 3 (3) | 1 (1) | 4 (4)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
COVID 19 (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Nasopharingitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Tonsilitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Venous Trombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Application site Swelling (General disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT04883632/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT04883632/SAP_001.pdf